CLINICAL TRIAL: NCT00741533
Title: Quality of Life in Thai Women Diagnosed Cervical Cancer at King Chulalongkorn Memorial Hospital
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dean,College of Public Health Sciences, Chulalongkorn University., College of Public Health Sciences, Chulalongkorn University.
Other Study IDs: CPHS-01
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Quality of Life; Cervical Cancer; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To study the quality of life of patients earlier diagnosed for cervical cancer and cervical intraepithelial neoplasia (CIN).

DETAILED DESCRIPTION:
In Thailand, age standardized incidence is 20.9 per 100,000 women-year. Treatment-related survival gain are experienced by side-effect that may reduce quality of life (QoL). We therefore, study the quality of life of patients earlier diagnosed for cervical cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Thai patients
* aged more than 15 years old.
* Diagnosed of cervical intraepithelial neoplasia (CIN) or cervical cancer with pathological confirmation. If she has more than one diseases, the most severe will be considered as diagnosis.
* Not suffered from confusion or reduced level of consciousness or unable to communicate.

Exclusion Criteria:

Ages: 15 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cervical intraepithelial neoplasia (CIN) or cervical cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Surasak Taneepanichskul, MD., Principal Investigator — College of Public Health Sciences, Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Patumwan, Bangkok, Thailand